CLINICAL TRIAL: NCT01345318
Title: A Multicenter Open-label Extension Study For Subjects Who Participated In Study B0151003 (Andante Ii)
Brief Title: B0151005 Open-Label Extension Study
Acronym: ANDANTE II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B0151005; 2011-000722-30 (EudraCT Number); ANDANTE II (Other: Alias Study Number)
Record Dates: First submitted 2011-04-28; First posted 2011-05-02 (Estimated); Results first posted 2017-03-20 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2017-01

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; safety; efficacy; pharmacokinetics; pharmacodynamics; Crohn's Disease Activity Index (CDAI)
MeSH Terms: conditions — Crohn Disease | interventions — PF-04236921

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open-label Treatment (Experimental)
  Interventions: Biological: PF-04236921

INTERVENTIONS:
Biological: PF-04236921 — Subjects entering this study will be given a 50 mg SC dose at baseline and then every 8 weeks through Week 40.
Biological: PF-04236921 — Dose escalation to 100 mg SC every 8 weeks will be allowed for subjects who have either not responded at Week 8 or have relapsed during the study.

SUMMARY:
This is a multi-center Phase 2, open label, safety extension study in subjects with moderate to severe CD who are anti-TNF inadequate responders. Subjects eligible for this study will have completed the 12-week induction period of study B0151003 and will be enrolled as either responders or non responders.

ELIGIBILITY:
Inclusion Criteria:

* Subjects previously enrolled in study B0151003 and completed the blinded 84 day (12 week) induction period.
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* Women of childbearing potential, who have sexual intercourse with a non surgically sterilized male partner, must agree and commit to the use highly effective methods of birth control from signing of the ICD through 26 weeks after the Final Study Evaluation or for 62 weeks from the last dose of investigational product for any subject who terminates early from this study.

Exclusion Criteria:

* Subjects that have completed Day 84 (Week 12) of study B0151003, and experienced serious event(s) related to the investigational product, an unstable medical condition, or any other reason, in the opinion of the investigator, would preclude entry or inclusion in this study.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate entry into this study.
* Received any prohibited treatment during study B0151003 that, in the opinion of the investigator, compromised the safety or efficacy of this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2011-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (127):
- United States (62):
  - Simon Medical Imaging, Scottsdale, Arizona
  - Digestive Health Research Unit, Scottsdale, Arizona
  - Adobe Clinical Research, LLC, Tucson, Arizona
  - Adobe Surgery Center, Tucson, Arizona
  - Rocky Mountain Gastroenterology Associates, Lakewood, Colorado
  - Rocky Mountain Gastroenterology, Littleton, Colorado
  - Rocky Mountain Clinical Research, LLC., Wheat Ridge, Colorado
  - Rocky Mountain Clinical Research, LLC, Wheat Ridge, Colorado
  - Medical Research Center of Connecticut, LLC, Hamden, Connecticut
  - Gastroenterology Consultants of Clearwater, Clearwater, Florida
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - Gastroenterology Associates, Crystal River, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - Suncoast Endoscopy Center, Inverness, Florida
  - International Clinical Research - US, LLC, Sanford, Florida
  - Atlanta Center for Gastroenterology, P.C., Decatur, Georgia
  - The Atlanta Center For Gastroenterology, Decatur, Georgia
  - Gastointestinal Specialists of Georgia, PC, Marietta, Georgia
  - Illinois Gastroenterology Group, LLC, Arlington Heights, Illinois
  - The University of Chicago Medical Center, Chicago, Illinois
  - NorthShore University Health System, Evanston, Illinois
  - University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - U of L Health Care Outpatient Center, Louisville, Kentucky
  - University of Louisville Hospital, Louisville, Kentucky
  - Digestive Disorders Associates, Annapolis, Maryland
  - Drgestive Disorders Associates, Annapolis, Maryland
  - East Valley Endoscopy, Grand Rapids, Michigan
  - Gastroenterology Associates of Western Michigan, Wyoming, Michigan
  - Metro Health Hospital Endoscopy Unit, Wyoming, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Huron Gastroenterology Associates, Ypsilanti, Michigan
  - Weill Cornell Medical College of Cornell University, New York, New York
  - Present, Chapman, Steinlauf and Marion, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - New York Presbyterian Hospital - Weill Cornell Medical College Investigational Pharmacy, New York, New York
  - Weill Cornell Imaging at New York Presbyterian Hospital, New York, New York
  - Weill Cornell Medical College of Cornell University-Greenberg, New York, New York
  - Arthur Asher Kombluth, MD PC, New York, New York
  - Oklahoma Foundation for Digestive Research, Oklahoma City, Oklahoma
  - Pharmacy: Wheeler and Stuckey, Inc., Oklahoma City, Oklahoma
  - Colonoscopy and X-rays: OU Physicians Building, Oklahoma City, Oklahoma
  - Hillcrest Medical Center, Tulsa, Oklahoma
  - Options Health Research, LLC, Tulsa, Oklahoma
  - Pittsburgh Gastroenterology Associates, Pittsburgh, Pennsylvania
  - Research Protocol Management Specialists, Pittsburgh, Pennsylvania
  - Gastro One, Germantown, Tennessee
  - Vanderbilt University Medical Center: IBD Clinic, Nashville, Tennessee
  - Vanderbilt University Medical Center-GI Research, Nashville, Tennessee
  - IBD Center-Vanderbilt University Medical Center, Nashville, Tennessee
  - Vanderbilt University Medical Center-IDS, Nashville, Tennessee
  - Professional Quality Research, Inc., Austin, Texas
  - Austin Gastroenterology, PA, Austin, Texas
  - Diagnostic Clinic Of Houston Pa, Houston, Texas
  - Diagnostic Clinic of Houston, PA, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - The University of TX Health Sci. Ctr at Houston, Houston, Texas
  - Texas Digestive Disease Consultants, Southlake, Texas
  - Clinical Pathologiy Laboratories, Inc, DBA DRL Labs, Tyler, Texas
  - Digestive Health Specialists of Tyler, Tyler, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - VC Medical Center Investigative Drug Service (IDS) [Ship Drug To], Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
- Australia (6):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Mater Health Services, South Brisbane, Queensland
  - Eastern Health, Box Hill Hospital, Box Hill, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - St. Vincent's Hospital, Fitzroy, Victoria
- Belgium (4):
  - CHU Saint-Pierre, Brussels
  - Chu St Pierre, Brussels
  - University Hospital Leuven, Campus Gasthuisberg, Leuven
  - H.-Hartziekenhuis Roeselare-Menen vzw, Roeselare
- Brazil (6):
  - Hospital Nossa Senhora das Gracas, Curitiba, Paraná
  - Setor de Cardiologia do Hospital Nossa Senhora das Gracas, Curitiba, Paraná
  - Setor de Endoscopia Digestiva do Hospital Nossa Senhora das Gracas, Curitiba, Paraná
  - Hospital Universitário Fraga Filho da UFRJ, Rio de Janeiro, Rio de Janeiro
  - Laboratório de Análises Clínicas do HUCFF/UFRJ, Rio de Janeiro, Rio de Janeiro
  - Hospital Israelita Albert Einstein, São Paulo, São Paulo
- Canada (4):
  - Heritage Medical Research Clinic - University of Calgary, Calgary, Alberta
  - London Health Science Centre - University Hospital, London, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Montreal General Hospital - McGill University Health Centre, Montreal, Quebec
- Czechia (5):
  - Hepato-Gastroenterologie HK, s.r.o. Poliklinika III, Hradec Králové
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni Nemocnice Kralovske Vinohrady, Prague
  - Institut klinicke a experimentalni mediciny, Prague
  - Krajska zdravotni, a.s., Ústí nad Labem
- Denmark (7):
  - Aarhus Universitetshospital, Aarhus Sygehus, Aarhus C
  - Rigshospitalet, Copenhagen
  - "Gastroenheden Herlev Hospital, Herlev
  - "Kirurgisk Afdeling 0143 Hilleroed Hospital, Hilleroed
  - Hvidovre Hospital, Hvidovre
  - Bispebjerg Hospital, Koebenhavn NV
  - Medicinsk Afdeling, Gastroenterologisk Sektion, Koege
- France (2):
  - Hopital Saint-Antoine - Service De Gastroenterologie, Paris, Cedex 12
  - Hopital Huriez CHRU de Lille, Lille
- Germany (4):
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Praxis Dr. Howaldt, Hamburg
  - Universitaetsklinikum Schleswig-Holstein, Kiel
  - Gastroenterologische Gemeinschaftspraxis Minden, Minden
- Hungary (4):
  - Pannonia Maganorvosi Centrum Kft., Budapest
  - Debreceni Egyetem Orvos- es Egeszsegtudomanyi Centrum, Debrecen
  - Szegedi Tudomanyegyetem altalanos Orvostudomanyi Kar / I. sz. Belgyogyaszati Klinika, Szeged
  - Clinfan Kft., Szekszárd
- Ireland (5):
  - National Virus Reference Laboratory, Dublin
  - Pathology, Haematology and Biochemistry Laboratories, St. Vincent's Healthcare Group, Dublin
  - Mater Misericordiae Hospital, Department of Clinical Chemistry and Clinical Haematology, Dublin
  - St. Vincents University Hospital, Dublin
  - University Hospital Galway, Galway
- Israel (6):
  - Digestive Disease Institute, Beith Vagan, Jerusalem
  - Institute of Gastroenterology, Haifa
  - Hadassah university Hospital (HUH) - Ein Karem, Hadassah Medical Organization (HMO), Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Beilinson Hospital, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (4):
  - Istituto Clinico Humanitas IRCCS, Rozzano, Milano
  - Azienda Ospedaliera - Universita di Padova, Padua
  - Universita Campus Biomedico UOC di Gastroenterologia, Roma
  - AOS San Camillo Forlanini, Rome
- New Zealand (2):
  - Shakespeare Specialist Group, Milford, Auckland
  - Waikato Hospital, Hamilton
- Universitaetsspital Zuerich, Zurich, Switzerland
- United Kingdom (5):
  - Addenbrookes Hospital, Cambridge
  - Glasgow Royal Infirmary, Glasgow
  - Barts Health NHS Trust-Royal London Hospital, London
  - Clinical Research Centre, London
  - St Bartholomew's Hospital (Barts Health NHS Trust), London

REFERENCES:
- [Derived] Danese S, Vermeire S, Hellstern P, Panaccione R, Rogler G, Fraser G, Kohn A, Desreumaux P, Leong RW, Comer GM, Cataldi F, Banerjee A, Maguire MK, Li C, Rath N, Beebe J, Schreiber S. Randomised trial and open-label extension study of an anti-interleukin-6 antibody in Crohn's disease (ANDANTE I and II). Gut. 2019 Jan;68(1):40-48. doi: 10.1136/gutjnl-2017-314562. Epub 2017 Dec 15. PMID 29247068
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0151005&StudyName=B0151005%20Open-Label%20Extension%20Study

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-04236921: All participants entering this study were given a 50 mg subcutaneous (SC) dose of PF-04236921 at baseline and then every 8 weeks through Week 40. The participants were on active treatment through Week 48. A one-time dose escalation to 100 mg was allowed, if participants experienced a clinical deterioration or unacceptably low level of response to study drug. Dose escalation was not allowed before Week 8.
Period: Overall Study
Arm/Group | PF-04236921
Started | 191
Completed | 111
Not Completed | 80
Not completed — Adverse Event | 16
Not completed — Lack of Efficacy | 17
Not completed — Lost to Follow-up | 2
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 41
Not completed — Other | 3

BASELINE CHARACTERISTICS:
Population: Included all participants who received at least 1 dose of study treatment during the study B0151005
Groups:
- PF-04236921: All participants entering this study were given a 50 mg SC dose of PF-04236921 at baseline and then every 8 weeks through Week 40. The participants were on active treatment through Week 48. A one-time dose escalation to 100 mg was allowed, if participants experienced a clinical deterioration or unacceptably low level of response to study drug. Dose escalation was not allowed before Week 8.
Arm/Group | PF-04236921
Number analyzed (Participants) | 191
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  FEMALE | 108
  MALE | 83

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With On-Treatment Treatment-Emergent Adverse Events (AEs), Serious Adverse Events (SAEs), and Discontinuations Due to AEs
Description: An AE was any untoward medical occurrence without regard to causality in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of death); persistent or significant disability/incapacity; congenital anomaly. Lack of efficacy was reported as an AE when it was associated with a SAE. An AE was considered treatment emergent if it started for the first time in a participant on or after the first day of active treatment, or the event started before the first day of active treatment but increased in severity during active treatment. AEs included both SAEs and non-serious AEs.
Time Frame: Baseline up to Week 48
Population: The safety analysis set was defined as all participants who received at least one dose of PF-04236921during the study.
Measure: Number; unit: participants
Arm/Group | PF-04236921
Number analyzed (Participants) | 191
participants
  Participants with AEs | 171
  Participants with SAEs | 58
  Participants discontinued due to AEs | 54

2. Primary Outcome: Percentage of Participants Developing Anti-Drug Antibodies (ADAs) and Neutralizing Antibodies (NAbs)
Description: Samples were analyzed using the semi-quantitative electrochemiluminescent (ECL) immunoassay method, a validated analytical method in compliance with sponsor's standard operating procedures. ADA positive is defined as ADA titer greater than or equal to (>=) 4.32. Any positive ADA sample was further tested for NAbs.
Time Frame: At Baseline and Weeks 8, 16, 24, 32, 40, 48, 56, 64, 72 and 76.
Population: The safety analysis set was defined as all participants who received at least one dose of PF-04236921during the study.
Measure: Number; unit: percentage of participants
Groups:
- PF-04236921: All participants entering this study were given a 50 mg SC dose of PF-04236921 at baseline and then every 8 weeks through Week 40. The participants were on active treatment through Week 48. A one-time dose escalation to 100 mg was allowed, if participants experienced clinical deterioration or unacceptably low level of response to study drug. Dose escalation was not allowed before Week 8.
Arm/Group | PF-04236921
Number analyzed (Participants) | 191
percentage of participants
  ADA positive | 0.52
  NAbs positive | 0.52

ADVERSE EVENTS:
Description: The same event might have appeared as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant might have experienced both a serious and non-serious event during the study.
Arm/Group | PF-04236921
Serious Adverse Events (participants affected / at risk) | 79/191
Other Adverse Events (participants affected / at risk) | 150/191
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | PF-04236921 (N=191)
Anaemia (Blood and lymphatic system disorders) | 1
Ulcerative keratitis (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain lower (Gastrointestinal disorders) | 1
Anal fistula (Gastrointestinal disorders) | 4
Anorectal disorder (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Crohn's disease (Gastrointestinal disorders) | 41
Dyspepsia (Gastrointestinal disorders) | 1
Enterovesical fistula (Gastrointestinal disorders) | 1
Fistula of small intestine (Gastrointestinal disorders) | 2
Gastritis erosive (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Large intestine perforation (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 2
Small intestinal obstruction (Gastrointestinal disorders) | 2
Small intestinal perforation (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 1
Cholangitis sclerosing (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 2
Cholecystitis chronic (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Abdominal abscess (Infections and infestations) | 4
Abscess (Infections and infestations) | 1
Anal abscess (Infections and infestations) | 1
Bartholin's abscess (Infections and infestations) | 1/108 — Percentages of gender specific events are calculated using the corresponding gender count as denominator.
Cellulitis (Infections and infestations) | 1
Cytomegalovirus infection (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 1
Groin abscess (Infections and infestations) | 1
Infectious colitis (Infections and infestations) | 1
Latent tuberculosis (Infections and infestations) | 1
Mesenteric abscess (Infections and infestations) | 1
Perirectal abscess (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Peritonsillar abscess (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Rectal abscess (Infections and infestations) | 1
Retroperitoneal abscess (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 2
Tooth abscess (Infections and infestations) | 1
Tuberculosis (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Viral upper respiratory tract infection (Infections and infestations) | 1
Anastomotic fistula (Injury, poisoning and procedural complications) | 1
Concussion (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Procedural complication (Injury, poisoning and procedural complications) | 1
Weight decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Multiple sclerosis relapse (Nervous system disorders) | 1
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 1/108 — Percentages of gender specific events are calculated using the corresponding gender count as denominator.
Calculus ureteric (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 2
Renal colic (Renal and urinary disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04236921 (N=191)
Anaemia (Blood and lymphatic system disorders) | 15
Abdominal pain (Gastrointestinal disorders) | 39
Crohn's disease (Gastrointestinal disorders) | 45
Diarrhoea (Gastrointestinal disorders) | 20
Nausea (Gastrointestinal disorders) | 21
Vomiting (Gastrointestinal disorders) | 22
Pyrexia (General disorders) | 14
Bronchitis (Infections and infestations) | 12
Gastroenteritis (Infections and infestations) | 11
Nasopharyngitis (Infections and infestations) | 31
Upper respiratory tract infection (Infections and infestations) | 11
Urinary tract infection (Infections and infestations) | 16
Arthralgia (Musculoskeletal and connective tissue disorders) | 23
Back pain (Musculoskeletal and connective tissue disorders) | 12
Headache (Nervous system disorders) | 23
Anxiety (Psychiatric disorders) | 10
Insomnia (Psychiatric disorders) | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 13
Erythema (Skin and subcutaneous tissue disorders) | 14
Rash (Skin and subcutaneous tissue disorders) | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.